CLINICAL TRIAL: NCT02360579
Title: A Phase 2, Multicenter Study to Assess the Efficacy and Safety of Autologous Tumor Infiltrating Lymphocytes (LN-144) for Treatment of Patients With Metastatic Melanoma
Brief Title: Study of Lifileucel (LN-144), Autologous Tumor Infiltrating Lymphocytes, in the Treatment of Patients With Metastatic Melanoma
Acronym: LN-144
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Iovance Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-144-01
Record Dates: First submitted 2015-02-03; First posted 2015-02-10 (Estimated); Results first posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Melanoma
Keywords: Autologous Adoptive Cell Transfer; Autologous Adoptive Cell Therapy; Cellular Immuno-therapy; Cell Therapy; Tumor Infiltrating Lymphocytes; TIL; LN-144; IL-2; Melanoma; Lifileucel
MeSH Terms: conditions — Melanoma | interventions — lifileucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Non-cryopreserved LN-144 (Gen 1 infusion product) (Closed)
  Interventions: Biological: Lifileucel
- Cohort 2 (Experimental): Cryopreserved lifileucel (LN-144) (Gen 2 infusion product) (Closed)
  Interventions: Biological: Lifileucel
- Cohort 3 (Experimental): Retreatment cohort: patients from Cohort 1, Cohort 2 or Cohort 4 may rescreen for a second TIL regimen therapy if they meet all Inclusion and Exclusion Criteria (except exclusion criterion b).
  Interventions: Biological: Lifileucel
- Cohort 4 (Experimental): Cryopreserved lifileucel (LN-144) (Gen 2 infusion product)
  Interventions: Biological: Lifileucel

INTERVENTIONS:
Biological: Lifileucel — A tumor sample is resected from each patient and cultured ex vivo to expand the population of tumor infiltrating lymphocytes. After lymphodepletion, patients are infused with lifileucel followed by IL-2.
  Other Names: LN - 144

SUMMARY:
Prospective, interventional multicenter study evaluating adoptive cell therapy (ACT) via infusion of LN-144 (autologous TIL) followed by interleukin 2 (IL-2) after a nonmyeloablative lymphodepletion (NMA LD) preconditioning regimen.

DETAILED DESCRIPTION:
Lifileucel is an autologous adoptive cell transfer therapy that utilizes a TIL manufacturing process, as originally developed by the NCI, for the treatment of patients with metastatic melanoma. The adoptive cell transfer therapy used in this study involves patients receiving a lymphocyte depleting preconditioning regimen, prior to infusion of autologous TIL, followed by the administration of a regimen of IL-2.

ELIGIBILITY:
Patients must meet all of the following inclusion criteria to be eligible for participation in the study:

Criteria for Inclusion:

1. Patients with unresectable or metastatic melanoma (Stage IIIc or Stage IV)
2. Patients must have progressed following ≥ one prior systemic therapy including a programmed cell death protein-1 (PD-1) blocking antibody; and if proto-oncogene B-Raf (BRAF) V600 mutation-positive, a BRAF inhibitor or BRAF inhibitor in combination with mitogen-activated extracellular signal-regulated kinase (MEK) inhibitor
3. At least one measurable target lesion, as defined by RECIST v1.1

   * Lesions in previously irradiated areas (or other local therapy) should not be selected as target lesions, unless treatment was ≥ 3 months prior to Screening, and there has been demonstrated disease progression in that particular lesion
4. At least one resectable lesion (or aggregate of lesions resected) of a minimum 1.5 cm in diameter post-resection to generate TIL; surgical removal with minimal morbidity (defined as any procedure for which expected hospitalization is ≤ 3 days)
5. Patients must be ≥ 18 years of age at the time of consent. Enrollment of patients > 70 years of age may be allowed after consultation with the Medical Monitor
6. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 and an estimated life expectancy of ≥ 3 months
7. In the opinion of the Investigator, patients must be able to complete all study-required procedures
8. Patients must have the following hematologic parameters:

   * Absolute neutrophil count (ANC) ≥ 1000/mm3
   * Hemoglobin (Hb) ≥ 9.0 g/dL
   * Platelet ≥ 100,000/mm3
9. Patients must have adequate organ function:

   * Serum alanine transaminase (ALT)/serum glutamic-pyruvic transaminase (SGPT) and aspartate transaminase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) ≤ 3 times the upper limit of normal (ULN); patients with liver metastasis ≤ 5 times ULN
   * Estimated creatinine clearance (eCrCl) ≥ 40 mL/min using the Cockcroft-Gault formula
   * Total bilirubin ≤ 2 mg/dL
   * Patients with Gilbert's syndrome must have a total bilirubin ≤ 3 mg/dL
10. Patients must have recovered from all prior therapy-related adverse events (AEs) to ≤ Grade 1 (per Common Terminology Criteria for Adverse Events [CTCAE] v4.03), except for alopecia or vitiligo, prior to Enrollment (tumor resection)

    * Patients with documented ≥ Grade 2 diarrhea or colitis as a result of previous treatment with immune checkpoint inhibitor(s) must have been asymptomatic for at least 6 months and/or had a normal colonoscopy post-immune checkpoint inhibitor treatment, by visual assessment, prior to tumor resection
11. Patients must have a washout period ≥ 28 days from prior anticancer therapy(ies) to the start of the planned NMA-LD preconditioning regimen:

    * Targeted therapy: MEK/BRAF or other targeted agent
    * Chemotherapy
    * Immunotherapy: anti-cytotoxic T lymphocyte-associated antigen 4 (CTLA-4)/anti-PD-1, other monoclonal antibody (mAb), or vaccine
    * Palliative radiation therapy is permitted so long as it does not involve lesions being selected for TIL, or as target or non-target lesions. Washout is not required if all related toxicities have resolved to ≤ Grade 1 as per CTCAE v4.03
12. Patients of childbearing potential or their partners of childbearing potential must be willing to take the appropriate precaution to avoid pregnancy or fathering a child for the duration of the study and practice an approved, highly effective method of birth control during treatment and for 12 months after receiving the last protocol-related therapy

    * Approved methods of birth control are as follows:
    * Combined (estrogen and progesterone containing) hormonal birth control associated with inhibition of ovulation: oral, intravaginal, transdermal
    * Progesterone-only hormonal birth control associated with inhibition of ovulation: oral, injectable, implantable
    * Intrauterine device (IUD)
    * Intrauterine hormone-releasing system (IUS)
    * Bilateral tubal occlusion
    * Vasectomized partner
    * True sexual abstinence when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (eg, calendar ovulation, symptothermal, post-ovulation methods) is not acceptable
13. Patients (or legally authorized representative) must have the ability to understand the requirements of the study, have provided written informed consent as evidenced by signature on an ICF approved by an Institutional Review Board/Independent Ethics Committee (IRB/IEC), and agree to abide by the study restrictions and return to the site for the required assessments, including the OS Follow-up Period
14. Patients have provided written authorization for use and disclosure of protected health information

Criteria for Exclusion:

Patients who meet any of the following criteria are not eligible for participation in this study:

1. Patients who have been shown to be BRAF mutation positive (V600), but have not received prior systemic therapy with a BRAF inhibitor alone or a BRAF inhibitor in combination with a MEK inhibitor
2. Patients who have received an organ allograft or prior cell transfer therapy
3. Patients with melanoma of uveal/ocular origin
4. Patients who have a history of hypersensitivity to any component or excipient of LN-144 or other study drugs:

   * NMA-LD preconditioning regimen (cyclophosphamide, mesna, and fludarabine)
   * Antibiotics (ABX) of the aminoglycoside group (ie, streptomycin, gentamicin); except those who are skin-test negative for gentamicin hypersensitivity
   * Any component of the LN-144 infusion product formulation including dimethyl sulfoxide (DMSO), human serum albumin (HSA), IL-2, and dextran-40
5. Patients with symptomatic and/or untreated brain metastases (of any size and any number)

   * Patients with definitively treated brain metastases may be considered for Enrollment, and must be stable for ≥ 14 days prior to beginning the NMA LD preconditioning regimen
6. Patients who are on chronic systemic steroid therapy for any reason
7. Patients who have active medical illness(es) that would pose increased risk for study participation, including: active systemic infections requiring systemic ABX, coagulation disorders, or other active major medical illnesses of the cardiovascular, respiratory, or immune system
8. Patients who have any form of primary immunodeficiency (such as severe combined immunodeficiency disease [SCID] and acquired immunodeficiency syndrome [AIDS])
9. Patients who have a left ventricular ejection fraction (LVEF) < 45% or New York Heart Association (NYHA) functional classification > Class 1

   * Patients ≥ 60 years of age and who have a history of ischemic heart disease, chest pain, or clinically significant atrial and/or ventricular arrhythmias must have a cardiac stress test. Patients with any irreversible wall movement abnormalities are excluded
10. Patients who have a documented forced expiratory volume in 1 second (FEV1) of ≤ 60%
11. Patients who have had another primary malignancy within the previous 3 years (with the exception of carcinoma in situ of the breast, cervix, or bladder; localized prostate cancer; and non-melanoma skin cancer that has been adequately treated)
12. Patients who have received a live or attenuated vaccine within 28 days of beginning the NMA-LD preconditioning regimen
13. Patients who are pregnant or breastfeeding
14. Patients whose cancer requires immediate attention or who would otherwise suffer a disadvantage by participating in this trial
15. Patients protected by the following constraints:

    * Hospitalized persons without consent or persons deprived of liberty because of a judiciary or administrative decision
    * Adult persons with a legal protection measure or persons who cannot express their consent
    * Patients in emergency situations who cannot consent to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2015-09-24 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iovance Biotherapeutics Medical Monitor, Study Chair — Iovance Biotherapeutics, Inc.
Locations (57):
- United States (23):
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - University of California Los Angeles - David Geffen School of Medicine - Westwood Rheumatology, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - University of Florida Health Cancer Center, Orlando, Florida
  - University of South Florida H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Indiana University, Indianapolis, Indiana
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - University of Minnesota, Masonic Cancer Center, Minneapolis, Minnesota
  - Atlantic Health System, Morristown, New Jersey
  - Rutgers University, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York University Langone Medical Center, New York, New York
  - Providence Cancer Center Oncology and Hematology Care Clinic, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- France (4):
  - Centre Léon Bérard, Lyon, Auvergne-Rhône-Alpes
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Hôpital Dupuytren, Limoges, Limousin
  - Gustave Roussy Cancer Campus, Villejuif, Île-de-France Region
- Germany (9):
  - Universitaetsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen (UKT) - Suedwestdeutschen Tumorzentrum - Zentrum für Neuroonkologie, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Klinikum Rechts der Isar der Technischen Universität München, München, Bavaria
  - Universitätsklinikum Carl Gustav Carus, Dresden, Saxony
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Universitätsklinikum Halle, Halle, Saxony-Anhalt
  - Universitätsklinikum Schleswig-Holstein - Campus Lübeck, Lübeck, Schleswig-Holstein
  - Universitätsklinikum Würzburg, Würzburg
- Szegedi Tudomanyegyetem Szent-Györgyi Albert Klinikai Központ, Szeged, Csongrád megye, Hungary
- Italy (5):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola, Forli-cesena
  - Centro di Riferimento Oncologico di Aviano, Aviano, Pordenone
  - Istituto di Candiolo - Fondazione del Piemonte per l'Oncologia, Candiolo, Torino
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli
- Spain (9):
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Institut Català d'Oncologia, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital 12 de Octubre, Madrid
  - HM Centro Integral Oncológico Clara Campal, Madrid
  - Hospital Universitario Quirónsalud Madrid, Madrid
  - Consorci Hospital General Universitari de València, Valencia
- Switzerland (2):
  - Inselspital, Bern
  - Centre Hospitalier Universitaire Vaudois Lausanne - Centre Pluridisciplinaire d'Oncologie, Lausanne
- United Kingdom (4):
  - Royal Marsden NHS Trust, London, England
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Addenbrooke's Hospital, Cambridge
  - Sarah Cannon Research Institute London, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chesney J, Lewis KD, Kluger H, Hamid O, Whitman E, Thomas S, Wermke M, Cusnir M, Domingo-Musibay E, Phan GQ, Kirkwood JM, Hassel JC, Orloff M, Larkin J, Weber J, Furness AJS, Khushalani NI, Medina T, Egger ME, Graf Finckenstein F, Jagasia M, Hari P, Sulur G, Shi W, Wu X, Sarnaik A. Efficacy and safety of lifileucel, a one-time autologous tumor-infiltrating lymphocyte (TIL) cell therapy, in patients with advanced melanoma after progression on immune checkpoint inhibitors and targeted therapies: pooled analysis of consecutive cohorts of the C-144-01 study. J Immunother Cancer. 2022 Dec;10(12):e005755. doi: 10.1136/jitc-2022-005755. PMID 36600653
- [Background] Medina T, Chesney JA, Kluger HM, Hamid O, Whitman ED, Cusnir M, Thomas SS, Wermke M, Domingo-Musibay E, Phan GQ, Kirkwood JM, Larkin J, Weber J, Graf Finckenstein F, Chou J, Gastman B, Wu X, Fiaz R, Sarnaik AA; C-144-01 Investigators. Long-Term Efficacy and Safety of Lifileucel Tumor-Infiltrating Lymphocyte Cell Therapy in Patients With Advanced Melanoma: A 5-Year Analysis of the C-144-01 Study. J Clin Oncol. 2025 Nov 20;43(33):3565-3572. doi: 10.1200/JCO-25-00765. Epub 2025 Jun 2. PMID 40454684
- [Background] Kluger H, Grigoleit GU, Thomas S, Domingo-Musibay E, Chesney JA, Sanmamed MF, Medina T, Ziemer M, Whitman E, Finckenstein FG, Gastman B, Chou J, Wu X, Sulur G, Fiaz R, Qi R, Sarnaik AA. Lifileucel tumor-infiltrating lymphocyte cell therapy in patients with unresectable or metastatic mucosal melanoma after disease progression on immune checkpoint inhibitors. Cancer Commun (Lond). 2025 Oct;45(10):1229-1234. doi: 10.1002/cac2.70050. Epub 2025 Jul 22. No abstract available. PMID 40693376
- [Derived] Sarnaik AA, Hamid O, Khushalani NI, Lewis KD, Medina T, Kluger HM, Thomas SS, Domingo-Musibay E, Pavlick AC, Whitman ED, Martin-Algarra S, Corrie P, Curti BD, Olah J, Lutzky J, Weber JS, Larkin JMG, Shi W, Takamura T, Jagasia M, Qin H, Wu X, Chartier C, Graf Finckenstein F, Fardis M, Kirkwood JM, Chesney JA. Lifileucel, a Tumor-Infiltrating Lymphocyte Therapy, in Metastatic Melanoma. J Clin Oncol. 2021 Aug 20;39(24):2656-2666. doi: 10.1200/JCO.21.00612. Epub 2021 May 12. PMID 33979178

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Cohorts 1, 2, 4 refers to the initial treatment. Cohort 3 patients had progressed following the initial treatment and then were retreated with a second TIL regimen. Data are captured in the retreatment period for Cohort 3.
Groups:
- Cohort 1: Non-cryopreserved LN-144 (Gen 1 infusion product) (Closed)
  A tumor sample is resected from each patient and cultured ex vivo to expand the population of tumor infiltrating lymphocytes. After lymphodepletion, patients are infused with lifileucel followed by IL-2.
- Cohort 3: Retreatment cohort: patients from Cohort 1, Cohort 2 or Cohort 4 may rescreen for a second TIL regimen therapy if they meet all Inclusion and Exclusion Criteria (except exclusion criterion b) (Closed)
  Lifileucel: A tumor sample is resected from each patient and cultured ex vivo to expand the population of tumor infiltrating lymphocytes. After lymphodepletion, patients are infused with lifileucel followed by IL-2.
- Cohort 4: Cryopreserved lifileucel (LN-144) (Gen 2 infusion product) (Closed)
  Lifileucel: A tumor sample is resected from each patient and cultured ex vivo to expand the population of tumor infiltrating lymphocytes. After lymphodepletion, patients are infused with lifileucel followed by IL-2.
Period: Initial
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 31 | 78 | 0 | 111
Patients Infused With TIL | 23 | 67 | 0 | 89
Completed (Completed refers to the number of patients who have received TIL and completed the study) | 0 | 14 | 0 | 14
Not Completed | 31 | 64 | 0 | 97
Not completed — Death | 16 | 49 | 0 | 71
Not completed — Lost to Follow-up | 0 | 4 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3
Not completed — Other | 7 | 0 | 0 | 0
Not completed — Did not receive TIL | 8 | 11 | 0 | 22
Period: Retreatment
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 0 | 0 (Cohort 3 patients had progressed following initial treatment in Cohorts 1, 2, 4 and then were retreated with a second TIL regimen. Data are captured in the retreatment period for Cohort 3) | 12 (Cohort 3 patients had progressed following initial treatment in Cohorts 1, 2, 4 and then were retreated with a second TIL regimen. Data are captured in the retreatment period for Cohort 3) | 0 (Cohort 3 patients had progressed following initial treatment in Cohorts 1, 2, 4 and then were retreated with a second TIL regimen. Data are captured in the retreatment period for Cohort 3)
Completed | 0 | 0 | 1 | 0
Not Completed | 0 | 0 | 11 | 0
Not completed — Death | 0 | 0 | 11 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set is defined as patients who received the lifileucel infusion. Cohort 3 patients had progressed following initial treatment in Cohorts 1, 2, 4 and then were retreated with a second TIL regimen. Data are captured in the retreatment period for Cohort 3
Groups:
- Cohort 3: Retreatment cohort: patients from Cohort 1, Cohort 2 or Cohort 4 may rescreen for a second TIL regimen therapy if they meet all Inclusion and Exclusion Criteria (except exclusion criterion b) (Closed)
- Cohort 4: Cryopreserved lifileucel (LN-144) (Gen 2 infusion product) (Closed)
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 23 | 67 | 12 | 89 | 191
Age, Categorical [Count of Participants; unit: Participants] — Population: Cohort 3 patients had progressed following initial treatment in Cohorts 1, 2, 4 and then were retreated with a second TIL regimen. Data prior to initial TIL treatment are presented in the retreatment period for Cohort 3
  Participants
    Initial Treatment: number analyzed (Participants) | 23 | 67 | 0 | 89 | 179
    Initial Treatment: <=18 years | 0 | 0 | 0 | 0 | 0
    Initial Treatment: Between 18 and 65 years | 21 | 53 | 0 | 66 | 140
    Initial Treatment: >=65 years | 2 | 14 | 0 | 23 | 39
    Retreatment: number analyzed (Participants) | 0 | 0 | 12 | 0 | 12
    Retreatment: <=18 years |  |  | 0 |  | 0
    Retreatment: Between 18 and 65 years |  |  | 11 |  | 11
    Retreatment: >=65 years |  |  | 1 |  | 1
Age, Continuous [Median (Full Range); unit: Years] — Population: Cohort 3 patients had progressed following initial treatment in Cohorts 1, 2, 4 and then were retreated with a second TIL regimen. Data prior to initial TIL treatment are presented in the retreatment period for Cohort 3
  Years
    Initial Treatment: number analyzed (Participants) | 23 | 67 | 0 | 89 | 179
    Initial Treatment | 52 [37 to 72] | 55 [20 to 79] |  | 58 [25 to 74] | 56 [20 to 79]
    Retreatment: number analyzed (Participants) | 0 | 0 | 12 | 0 | 12
    Retreatment |  |  | 52 [29 to 66] |  | 52 [29 to 66]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Cohort 3 patients had progressed following initial treatment in Cohorts 1, 2, 4 and then were retreated with a second TIL regimen. Data prior to initial TIL treatment are presented in the retreatment period for Cohort 3
  Participants
    Initial Treatment: number analyzed (Participants) | 23 | 67 | 0 | 89 | 179
    Initial Treatment: Female | 12 | 28 | 0 | 44 | 84
    Initial Treatment: Male | 11 | 39 | 0 | 45 | 95
    Retreatment: number analyzed (Participants) | 0 | 0 | 12 | 0 | 12
    Retreatment: Female | 0 | 0 | 3 | 0 | 3
    Retreatment: Male | 0 | 0 | 9 | 0 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Cohort 3 patients had progressed following initial treatment in Cohorts 1, 2, 4 and then were retreated with a second TIL regimen. Data prior to initial TIL treatment are presented in the retreatment period for Cohort 3
  Participants
    Initial Treatment: number analyzed (Participants) | 23 | 67 | 0 | 89 | 179
    Initial Treatment: Hispanic or Latino | 2 | 5 | 0 | 3 | 10
    Initial Treatment: Not Hispanic or Latino | 21 | 55 | 0 | 85 | 161
    Initial Treatment: Unknown or Not Reported | 0 | 7 | 0 | 1 | 8
    Retreatment: number analyzed (Participants) | 0 | 0 | 12 | 0 | 12
    Retreatment: Hispanic or Latino | 0 | 0 | 1 | 0 | 1
    Retreatment: Not Hispanic or Latino | 0 | 0 | 10 | 0 | 10
    Retreatment: Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Cohort 3 patients had progressed following initial treatment in Cohorts 1, 2, 4 and then were retreated with a second TIL regimen. Data prior to initial TIL treatment are presented in the retreatment period for Cohort 3
  Participants
    Initial Treatment: number analyzed (Participants) | 23 | 67 | 0 | 89 | 179
    Initial Treatment: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Initial Treatment: Asian | 0 | 2 | 0 | 1 | 3
    Initial Treatment: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Initial Treatment: Black or African American | 0 | 1 | 0 | 2 | 3
    Initial Treatment: White | 23 | 64 | 0 | 85 | 172
    Initial Treatment: More than one race | 0 | 0 | 0 | 0 | 0
    Initial Treatment: Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
    Retreatment: number analyzed (Participants) | 0 | 0 | 12 | 0 | 12
    Retreatment: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Retreatment: Asian | 0 | 0 | 0 | 0 | 0
    Retreatment: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Retreatment: Black or African American | 0 | 0 | 2 | 0 | 2
    Retreatment: White | 0 | 0 | 9 | 0 | 9
    Retreatment: More than one race | 0 | 0 | 0 | 0 | 0
    Retreatment: Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants] — Population: Cohort 3 patients had progressed following initial treatment in Cohorts 1, 2, 4 and then were retreated with a second TIL regimen. Data prior to initial TIL treatment are presented in the retreatment period for Cohort 3
  Participants
    United States: number analyzed (Participants) | 23 | 67 | 0 | 89 | 179
    United States | 23 | 56 | 0 | 55 | 134
    France: number analyzed (Participants) | 23 | 67 | 0 | 89 | 179
    France | 0 | 2 | 0 | 1 | 3
    Germany: number analyzed (Participants) | 23 | 67 | 0 | 89 | 179
    Germany | 0 | 0 | 0 | 19 | 19
    Hungary: number analyzed (Participants) | 23 | 67 | 0 | 89 | 179
    Hungary | 0 | 2 | 0 | 0 | 2
    Spain: number analyzed (Participants) | 23 | 67 | 0 | 89 | 179
    Spain | 0 | 3 | 0 | 10 | 13
    Switzerland: number analyzed (Participants) | 23 | 67 | 0 | 89 | 179
    Switzerland | 0 | 1 | 0 | 0 | 1
    United Kingdom: number analyzed (Participants) | 23 | 67 | 0 | 89 | 179
    United Kingdom | 0 | 3 | 0 | 4 | 7
Region of Enrollment [Count of Participants; unit: Participants] — Region of enrollment for retreatment Population: This is the region of enrollment for retreatment
  Participants
    number analyzed (Participants) | 0 | 0 | 12 | 0 | 12
    United States | 0 | 0 | 8 | 0 | 8
    France | 0 | 0 | 1 | 0 | 1
    Germany | 0 | 0 | 2 | 0 | 2
    United Kingdom | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Disease Assessment for Objective Response Rate
Description: Evaluate the efficacy of LN-144 in patients with unresectable or metastatic melanoma using the objective response rate (ORR), as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 for Cohorts 1 & 3 and as assessed by Independent Review Committee (IRC) per RECIST Version 1.1 for Cohorts 2 & 4
Time Frame: Every 6 weeks for 6 months, then every 3 months for a maximum of 60 months
Population: The Full Analysis Set is defined as patients who received the lifileucel infusion that met product manufacturing specifications. Cohort 3 patients had progressed following initial treatment in Cohorts 1, 2, 4 and then were retreated with a second TIL regimen.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 20 | 66 | 10 | 87
Participants | 4 | 23 | 1 | 25

2. Secondary Outcome: Disease Assessment for Duration of Response
Description: Evaluate the efficacy endpoints of duration of response (DOR) by the IRC for Cohorts 2 & 4 and by the investigator for Cohort 1 per RECIST v1.1
Time Frame: Every 6 weeks for 6 months, then every 3 months for a maximum of 60 months
Population: The Full Analysis Set is defined as patients who received the lifileucel infusion that met product manufacturing specifications. Due to the small number of patients this outcome measure was not analyzed for Cohort 3 per the statistical analysis plan.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Cohort 2; Cohort 4: Cryopreserved lifileucel (LN-144) (Gen 2 infusion product)
- Cohort 1: Non-cryopreserved LN-144 (Gen 1 infusion product)
Arm/Group | Cohort 2 | Cohort 4 | Cohort 1
Number analyzed (Participants) | 23 | 25 | 4
months | NA [NA to NA] — Insufficient number of participants with events, therefore the Median and 95% Confidence Interval were not reached | 10.4 [4.1 to 26.2] | NA [3.0 to NA] — Insufficient number of participants with events, therefore the Median and 95% Confidence Interval were not reached

3. Secondary Outcome: Disease Assessment for Disease Control Rate
Description: Evaluate the efficacy endpoints of disease control rate (DCR) by the IRC for Cohorts 2 & 4 and by the investigator for Cohort 1 per RECIST v1.1
Time Frame: Every 6 weeks for 6 months, then every 3 months for a maximum of 60 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2 | Cohort 4 | Cohort 1
Number analyzed (Participants) | 66 | 87 | 20
Participants | 48 | 72 | 12

4. Secondary Outcome: Disease Assessment for Progression-Free Survival
Description: Evaluate the efficacy endpoints of Progression-Free Survival by the IRC for Cohorts 2 & 4 and by the investigator for Cohort 1 per RECIST v1.1
Time Frame: Every 6 weeks for 6 months, then every 3 months for a maximum of 60 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 2 | Cohort 4 | Cohort 1
Number analyzed (Participants) | 66 | 87 | 20
months | 4.1 [2.8 to 8.4] | 3.9 [2.8 to 4.9] | 2.6 [1.4 to 4.2]

5. Secondary Outcome: Overall Survival
Description: Evaluate overall survival (OS)
Time Frame: Until death or up to 60 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 2 | Cohort 4 | Cohort 1
Number analyzed (Participants) | 66 | 87 | 20
months | 15.6 [11.0 to 23.3] | 12.7 [8.3 to 17.8] | 12.9 [5.3 to 26.1]

ADVERSE EVENTS:
Time Frame: From enrollment to end of follow-up (up to 5 years)
Description: Treatment-emergent adverse events (TEAEs), clinical laboratory data assessments, serious adverse events (SAEs), and adverse events (AEs) were collected and evaluated for the duration of the study until resolution or permanent sequelae. The Safety Analysis Set is defined as patients who have received TIL infusion.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 18/23 | 49/67 | 11/12 | 71/89
Serious Adverse Events (participants affected / at risk) | 9/23 | 23/67 | 2/12 | 31/89
Other Adverse Events (participants affected / at risk) | 23/23 | 67/67 | 12/12 | 89/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=23) | Cohort 2 (N=67) | Cohort 3 (N=12) | Cohort 4 (N=89)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 6 | 0 | 2
Neutropenia [1] (Blood and lymphatic system disorders) | 1 | 1 | 1 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia [2] (Blood and lymphatic system disorders) | 3 | 4 | 2 | 3
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Uveitis (Eye disorders) | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 2 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 2 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 2
Sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 2 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 1
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 0 | 2
Oliguria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 0 | 2
Embolism (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 2
Shock (Vascular disorders) | 0 | 0 | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=23) | Cohort 2 (N=67) | Cohort 3 (N=12) | Cohort 4 (N=89)
Anaemia (Blood and lymphatic system disorders) | 18 | 46 | 11 | 54
Febrile neutropenia (Blood and lymphatic system disorders) | 11 | 30 | 5 | 27
Leukopenia [1] (Blood and lymphatic system disorders) | 12 | 28 | 2 | 29
Lymphopenia [2] (Blood and lymphatic system disorders) | 6 | 23 | 3 | 28
Neutropenia [3] (Blood and lymphatic system disorders) | 11 | 37 | 5 | 30
Normocytic anaemia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 4
Pancytopenia (Blood and lymphatic system disorders) | 1 | 5 | 0 | 4
Thrombocytopenia [4] (Blood and lymphatic system disorders) | 17 | 60 | 10 | 72
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 1 | 3
Sinus tachycardia (Cardiac disorders) | 6 | 10 | 1 | 13
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 3 | 1 | 1
Tachycardia (Cardiac disorders) | 3 | 23 | 6 | 22
Deafness bilateral (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 2 | 0 | 0 | 1
Uveitis (Eye disorders) | 0 | 3 | 1 | 2
Vision blurred (Eye disorders) | 0 | 4 | 0 | 4
Abdominal distension (Gastrointestinal disorders) | 2 | 1 | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 4 | 1 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 6 | 0 | 2
Constipation (Gastrointestinal disorders) | 4 | 13 | 1 | 7
Diarrhoea (Gastrointestinal disorders) | 9 | 19 | 5 | 29
Dry mouth (Gastrointestinal disorders) | 1 | 5 | 0 | 8
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 0 | 1
Nausea (Gastrointestinal disorders) | 13 | 16 | 2 | 21
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 4
Vomiting (Gastrointestinal disorders) | 9 | 14 | 2 | 20
Asthenia (General disorders) | 2 | 8 | 0 | 14
Chills (General disorders) | 15 | 52 | 9 | 64
Fatigue (General disorders) | 8 | 26 | 1 | 25
Malaise (General disorders) | 2 | 4 | 0 | 5
Mucosal inflammation (General disorders) | 0 | 4 | 0 | 4
Non-cardiac chest pain (General disorders) | 2 | 2 | 0 | 2
Oedema (General disorders) | 1 | 1 | 1 | 8
Oedema peripheral (General disorders) | 8 | 17 | 3 | 15
Pain (General disorders) | 1 | 1 | 1 | 2
Pyrexia (General disorders) | 9 | 39 | 6 | 42
Cytokine release syndrome (Immune system disorders) | 0 | 1 | 1 | 4
Hypersensitivity (Immune system disorders) | 2 | 0 | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 5
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 7 | 15 | 4 | 13
Aspartate aminotransferase increased (Investigations) | 5 | 19 | 4 | 13
Blood alkaline phosphatase increased (Investigations) | 6 | 14 | 2 | 9
Blood bilirubin increased (Investigations) | 3 | 5 | 1 | 7
Blood creatine phosphokinase increased (Investigations) | 0 | 5 | 1 | 5
Blood creatinine increased (Investigations) | 1 | 5 | 2 | 9
Breath sounds abnormal (Investigations) | 0 | 1 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 1 | 4
International normalised ratio increased (Investigations) | 0 | 1 | 1 | 2
Urine output decreased (Investigations) | 0 | 4 | 0 | 1
Weight decreased (Investigations) | 3 | 9 | 3 | 8
Weight increased (Investigations) | 1 | 16 | 1 | 10
Decreased appetite (Metabolism and nutrition disorders) | 7 | 19 | 2 | 11
Dehydration (Metabolism and nutrition disorders) | 6 | 5 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 | 14 | 0 | 14
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 16 | 1 | 13
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 17 | 3 | 26
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 16 | 4 | 15
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 11 | 2 | 8
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 30 | 5 | 28
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 6 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 9 | 2 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 5
Dizziness (Nervous system disorders) | 2 | 6 | 1 | 5
Headache (Nervous system disorders) | 3 | 8 | 0 | 12
Lethargy (Nervous system disorders) | 0 | 1 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 2 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 5 | 0 | 9
Confusional state (Psychiatric disorders) | 1 | 9 | 1 | 5
Delirium (Psychiatric disorders) | 0 | 4 | 0 | 5
Insomnia (Psychiatric disorders) | 2 | 6 | 1 | 7
Acute kidney injury (Renal and urinary disorders) | 1 | 6 | 0 | 9
Haematuria (Renal and urinary disorders) | 0 | 5 | 1 | 4
Oliguria (Renal and urinary disorders) | 0 | 3 | 0 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 13 | 0 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 14 | 0 | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 16 | 2 | 18
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 0 | 8
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 9
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 10
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 0 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 19 | 0 | 19
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 4 | 0 | 4
Erythema (Skin and subcutaneous tissue disorders) | 4 | 4 | 0 | 3
Petechiae (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 13 | 1 | 11
Rash (Skin and subcutaneous tissue disorders) | 0 | 16 | 3 | 23
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 14 | 1 | 10
Vitiligo (Skin and subcutaneous tissue disorders) | 3 | 6 | 0 | 3
Capillary leak syndrome (Vascular disorders) | 0 | 8 | 2 | 10
Flushing (Vascular disorders) | 2 | 4 | 1 | 4
Hypertension (Vascular disorders) | 4 | 9 | 2 | 17
Hypotension (Vascular disorders) | 7 | 24 | 5 | 27
Thrombophlebitis (Vascular disorders) | 0 | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (8):
  • Study Protocol: Protocol V9.0 (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/79/NCT02360579/Prot_000.pdf
  • Study Protocol: Protocol V8.0 (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT02360579/Prot_001.pdf
  • Study Protocol: Protocol V3.0 (2015-07-16): https://cdn.clinicaltrials.gov/large-docs/79/NCT02360579/Prot_002.pdf
  • Study Protocol: Protocol V4.0 (2016-07-18): https://cdn.clinicaltrials.gov/large-docs/79/NCT02360579/Prot_003.pdf
  • Study Protocol: Protocol V5.0 (Incorporating Amendments 1-4) (2017-02-04): https://cdn.clinicaltrials.gov/large-docs/79/NCT02360579/Prot_004.pdf
  • Study Protocol: Protocol V7.0_(Incorporating Amendments 1 through 6) (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/79/NCT02360579/Prot_005.pdf
  • Study Protocol: Protocol V6.0 (Incorporating Amendments 1-5) (2017-05-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT02360579/Prot_006.pdf
  • Statistical Analysis Plan (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/79/NCT02360579/SAP_007.pdf